CLINICAL TRIAL: NCT00027560
Title: Phase II Trial Of Non-Myeloablative Regimen Combining Melphalan, Fludarabine, And Anti-CD52 Monoclonal Antibody (CAMPATH-1H) Followed By An Unmodified Hematopoietic Cell Transplant From An HLA Compatible Related Or Unrelated Donor For Treatment Of Lymphohematopoietic Malignancies
Brief Title: Melphalan, Fludarabine, and Alemtuzumab Followed by Peripheral Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-092; MSKCC-01092; NCI-G01-2028
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; Waldenström macroglobulinemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Alemtuzumab; Cyclosporine; fludarabine phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES (Experimental): This is a stratified single-armed phase II study designed to investigate the safety and efficacy of hematopoietic cell allografts administered after nonmyeloablative cytoreduction.
  Interventions: Biological: alemtuzumab; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: melphalan; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: alemtuzumab — Consenting individuals will receive pretransplant immunosuppressive cytoreduction, which will consist of 4 days of Campath-1H, 5 days of fludarabine, and two days of melphalan. All therapy should be completed approximately 24-36 hours before administration of the primary allograft.
  Campath-1H (20mg/dose/day) will be administered for each of four days from day -8 to day -5, inclusive. Each dose will be infused intravenously over 8 hours.
  Other Names: Campath
Drug: cyclosporine — Patients will be treated with Cyclosporine as prophylaxis against GvHD. Cyclosporine will be initiated at least 1 day prior to transplant at a dose of 1.5 mg / kg IV q12h (3 mg / kg / day = total daily dose). Dose will thereafter be adjusted to maintain a trough serum level of 200-300 ng /ml. Cyclosporine will be administered intravenously until the patient tolerates full alimentation, at which time conversion to oral dosing to sustain therapeutic levels will be initiated according to standard BMT service guidelines.
Drug: fludarabine phosphate — Fludarabine, 25mg/m2/d will be administered for each of five days from day -8 to day -4, inclusive. Each dose will be infused intravenously over 30 minutes.
Drug: melphalan — Melphalan will be administered intravenously over 30 minutes on each of two days from day -3 to day -2, inclusive. The dose for recipients of HLA-matched related grafts will be 50 mg/m2/day x 2. The dose for recipients of HLA-matched unrelated and HLA-single allele disparate related or unrelated marrow or PBSC transplants will be 70 mg/m2/day x 2.
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as melphalan and fludarabine, and a monoclonal antibody, such as alemtuzumab, before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well fludarabine, melphalan, alemtuzumab, and peripheral stem cell transplant work in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Overall survival-12 months

Overall survival-24 months

Acute Graft-versus-Host Disease Matched Related patients-up to 4 months post transplant

Acute Graft-versus-Host Disease Unrelated and Mismatched related patients- up to 4 months post transplant

Chronic Graft-versus-Host Disease Matched Related patients- up to 2 years post transplant

Chronic Graft-versus-host disease Unrelated and Mismatched related patients- up to 2 years post transplant

* OUTLINE: Patients are stratified according to donor type (HLA-matched related vs HLA-matched unrelated, single HLA-allele disparate related, or unmatched) (HLA-mismatched related or matched unrelated donor stratum closed to accrual as of 1/11/06).

Patients receive a nonmyeloablative regimen comprising alemtuzumab IV over 8 hours on days -8 to -5, fludarabine IV over 30 minutes on days -8 to -4, and melphalan IV over 30 minutes on days -3 and -2. Allogeneic peripheral blood stem cells or bone marrow is infused on day 0.

Patients receive graft-versus host disease prophylaxis comprising cyclosporine IV every 12 hours beginning on day -1 and continuing orally as tolerated until day 100.

Patients are followed every 6 weeks for 6 months, every 3 months for 6 months, every 3-6 months for 1 year, and then annually thereafter or as clinically indicated.

PROJECTED ACCRUAL: A maximum of 50 patients (25 HLA-matched related and 25 HLA-mismatched related or matched unrelated) will be accrued for this study within 2 years (HLA-mismatched related or matched unrelated donor stratum closed to accrual as of 1/11/06).

ELIGIBILITY:
INCLUSION CRITERIA:

* Disease criteria: This trial is primarily designed for: 1) patients with relapsed or primary refractory non-Hodgkin's lymphoma, 2) chemosensitive relapsed or refractory acute and chronic lymphocytic leukemias, 3) relapsed or primary refractory Hodgkin's Disease, or advanced (Durie-Salmon stage II or III) multiple myeloma, advanced Waldenstrom macroglobulinemia, who, by virtue of advanced age, intensity of prior radiation and/or chemotherapy, history of prior toxicity associated with chemo/radiotherapy or existing organ dysfunction, would be at undue risk of regimen associated mortality if transplanted according to protocols involving myeloablative conditioning regimens.
* Patients with aggressive NHL histologies must have chemo/radiosensitive disease, or have non-progressive disease, or have stable disease on therapy, and be ineligible for an autologous HSC transplant because of disease in the marrow.
* Patients with chronic myeloid leukemia and high risk forms of acute myelogenous leukemia or myelodysplastic syndromes are also eligible in the absence of an alternative active higher priority allogeneic transplant protocol for which they are eligible.
* Age criteria: Patients may be up to 70 years of age. There is no lower age threshold. Patients above the age of 70 may also participate, after evaluation and approval by the BMT Service attendings.
* Absence of active or uncontrolled bacterial, viral, or fungal infection that would contraindicate the use of myelosuppressive chemotherapy.
* Patients must have a healthy HLA-compatible donor, either a matched or single HLA allele disparate related donor or a similarly compatible unrelated donor recruited through the National Marrow Donor Program. Related donors must be willing to participate as research subjects and be willing to receive G-CSF to mobilize PBPC and undergo leukapheresis to donate PBSC. Unrelated donors identified by the NMDP may elect to donate either PBSC after treatment with G-CSF, or bone marrow. These unrelated donors will provide informed consent and their PBSC or bone marrow donations will be obtained at a qualified donor center participating in the NMDP.
* Each patient must be willing to participate as a research subject and must sign an informed consent form after discussion of the nature and risks of the study prior to entering the protocol. Parents or legal guardians of patients who are minors will sign the consent form for these patients after discussion of the nature and risks of the study.

EXCLUSION CRITERIA:

* Female patients who are pregnant or lactating.
* Active or uncontrolled viral (including HIV-1), bacterial or fungal infection.
* Severe renal insufficiency (creatinine >2.0 or creatinine clearance < 30mL/minute)
* Severe hepatic dysfunction, as defined by: total bilirubin greater than 2.5 mg/dL and AST and ALT >3xnl, unless the liver is involved with disease.
* Severe cardiac insufficiency, defined as a resting left ventricular ejection of less than 30% as measured by echocardiography or radionuclide cardiac angiography. Patients on cardiac medications for congestive heart failure are eligible, as long as their LVEF is greater than 30% on medication.
* Severe pulmonary insufficiency, as defined by an adjusted diffusing capacity of less than 40% of predicted value.
* Karnofsky or Lansky score <40%

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2001-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo R. Castro-Malaspina, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 07/31/2001 Protocol Closed to Accrual 05/23/2006 Primary Completion Date 04/14/2009 Recruitment Location is medical clinic
Pre-assignment Details: Enrolled participants receive preparative cytoreduction prior to transplant.
Period: Overall Study
Arm/Group | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES
Started | 51
Completed | 50
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 46
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 42.9 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 12 months post transplant
Population: Population is defined as all participants who received transplant as per protocol.
Measure: Number; unit: participants
Arm/Group | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES
Number analyzed (Participants) | 50
participants | 37

2. Primary Outcome: Overall Survival
Time Frame: 24 months post transplant
Population: Population is defined as all participants who received transplant as per protocol.
Measure: Number; unit: participants
Arm/Group | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES
Number analyzed (Participants) | 50
participants | 30

3. Primary Outcome: Acute Graft-versus-Host Disease Matched Related Patients
Description: Grade III-IV Acute Graft-versus-Host Disease
Time Frame: up to 4 months post transplant
Population: The number of matched related patients was analyzed as per protocol.
Measure: Number; unit: participants
Arm/Group | Matched Related Patients
Number analyzed (Participants) | 25
participants | 1

4. Secondary Outcome: Acute Graft-versus-Host Disease Unrelated and Mismatched Related Patients
Description: Grade III-IV Acute Graft-versus-Host Disease
Time Frame: up to 4 months post transplant
Population: The number of unrelated and mismatched patients was analyzed as per protocol.
Measure: Number; unit: participants
Arm/Group | Unrelated and Mismatched Related Patients
Number analyzed (Participants) | 25
participants | 3

5. Secondary Outcome: Extensive Chronic Graft-versus-Host Disease Matched Related Patients
Time Frame: up to 2 years post transplant
Population: The number of matched related patients was analyzed as per protocol.
Measure: Number; unit: participants
Arm/Group | Matched Related Patients
Number analyzed (Participants) | 25
participants | 0

6. Secondary Outcome: Extensive Chronic Graft-versus-Host Disease Unrelated and Mismatched Related Patients
Time Frame: up to 2 years post transplant
Population: The number of unrelated and mismatched patients was analyzed as per protocol.
Measure: Number; unit: participants
Arm/Group | Unrelated and Mismatched Related Patients
Number analyzed (Participants) | 25
participants | 2

ADVERSE EVENTS:
Time Frame: Weekly during the first 3 months post transplant, every 6 weeks during months 3-6 and then 3 month intervals for 1 year post transplant
Arm/Group | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 43/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES (N=50)
Infection with grade 3/4 neut (Infections and infestations) | 1 (1)
Infection w.out neutropenia (Infections and infestations) | 1 (1)
Constitut symp, other (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TREATMENT OF LYMPHOHEMATOPOIETIC MALIGNANCIES (N=50)
SGOT (AST) (Hepatobiliary disorders) | 8
Bilirubin increased (Hepatobiliary disorders) | 12
Stomatitis/BMT (Gastrointestinal disorders) | 9
Alkaline phosphatase (Hepatobiliary disorders) | 8
Creatinine increased (Metabolism and nutrition disorders) | 32
Hyperglycemia (Blood and lymphatic system disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13
Transfusion (PLT/BMT) (Blood and lymphatic system disorders) | 9
SGPT (ALT) (Hepatobiliary disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes